CLINICAL TRIAL: NCT02112838
Title: A Phase 2, Multi-Center, Randomised, Double-Blind, Ascending-Dose, Placebo-Controlled Clinical Study to Assess the Safety and Efficacy of Fostamatinib in the Treatment of IgA Nephropathy
Brief Title: Safety and Efficacy Study of Fostamatinib to Treat Immunoglobin A (IgA) Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-935788-050; 2014-000331-16 (EudraCT Number)
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Results first posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: IGA Nephropathy
Keywords: IGA Glomerulonephritis; Nephritis, IGA Type
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — fostamatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fostamatinib 150 mg (Active Comparator): Fostamatinib 150 milligram (mg) tablet twice daily by mouth, over the course of 24 weeks
  Interventions: Drug: Fostamatinib 150 mg
- Fostamatinib 100 mg (Active Comparator): Fostamatinib 100 mg tablet twice daily by mouth, over the course of 24 weeks
  Interventions: Drug: Fostamatinib 100 mg
- Placebo (Placebo Comparator): Placebo tablet twice daily by mouth, over the course of 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fostamatinib 150 mg — Fostamatinib 150 milligram (mg) tablet twice daily by mouth, over the course of 24 weeks
  Other Names: R935788; R788
  Arms: Fostamatinib 150 mg
Drug: Fostamatinib 100 mg — Fostamatinib 100 mg tablet twice daily by mouth, over the course of 24 weeks
  Other Names: R935788; R788
  Arms: Fostamatinib 100 mg
Drug: Placebo — Placebo tablet twice daily by mouth, over the course of 24 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether fostamatinib is safe and effective in the treatment of IgA Nephropathy

ELIGIBILITY:
Inclusion Criteria:

* Renal biopsy findings consistent with IgA nephropathy
* Treatment with an Angiotensin Converting Enzyme inhibitor (ACEi) and/or an Angiotensin II Receptor Blocker (ARB) for at least 90 days at the maximum approved (or tolerated) dose
* Proteinuria > 1 gm/day at diagnosis of IgA nephropathy and Proteinuria > 0.50 gm/day at the second Screening Visit
* Blood pressure controlled to ≤ 130/80 with angiotensin blockade with or without other anti-hypertensive agents

Exclusion Criteria:

* Recent use of cyclophosphamide, mycophenolate mofetil, azathioprine, or Rituximab.
* Use of > 15 mg/day prednisone (or other corticosteroid equivalent).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-10; Primary Completion 2018-03-23 (Actual); Study Completion 2018-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rigel Pharmaceuticals, Inc., Study Director — Rigel Pharmaceuticals,Inc.
Locations (20):
- United States (4):
  - Stanford University Medical, Palo Alto, California
  - Nephrology Associates PC, University Hospital, Professional Center 1, Augusta, Georgia
  - Ohio State University, Columbus, Ohio
  - Southeast Renal Research Institute, Chattanooga, Tennessee
- Austria (2):
  - Medical University of Graz, Graz, Styria
  - Medical University Vienna, Nephrology, Vienna
- Germany (4):
  - Medical University of Heidelberg, Heidelberg, Baden-Wurtemberberg
  - Klinikum der Universität München, Munich, Bavaria
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden, Saxony
  - Medical University of Jena, Jena, Thuringia
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong, Sha Tin
  - Queen Mary Hospital, Hong Kong
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - School of Medicine, Chang Gung University, Chang Gung Memorial Hospital, Taoyuan District
- United Kingdom (6):
  - Addenbrookes Hospital, Cambridge
  - Cardiff University, Cardiff
  - Leicester General Hospital, Leicester
  - Royal Free Hospital, London
  - Hammersmith Hospital, London
  - Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prendecki M, Gulati K, Turner-Stokes T, Bhangal G, Chiappo D, Woollard K, Cook HT, Tam FW, Roufosse C, Pusey CD, McAdoo SP. Characterisation of an enhanced preclinical model of experimental MPO-ANCA autoimmune vasculitis. J Pathol. 2021 Oct;255(2):107-119. doi: 10.1002/path.5746. Epub 2021 Jul 23. PMID 34124781
- [Derived] McAdoo S, Tam FWK. Role of the Spleen Tyrosine Kinase Pathway in Driving Inflammation in IgA Nephropathy. Semin Nephrol. 2018 Sep;38(5):496-503. doi: 10.1016/j.semnephrol.2018.05.019. PMID 30177021
- [Derived] Yeo SC, Liew A, Barratt J. Emerging therapies in immunoglobulin A nephropathy. Nephrology (Carlton). 2015 Nov;20(11):788-800. doi: 10.1111/nep.12527. PMID 26032537

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fostamatinib 150 mg | Fostamatinib 100 mg | Placebo
Started | 25 | 26 | 25
Completed | 20 | 24 | 24
Not Completed | 5 | 2 | 1

BASELINE CHARACTERISTICS:
Population: the 76 subjects who were randomized and received at least 1 dose of the blinded study drug comprised the ITT Population, the Safety Population, and the PK Population. Paired biopsies with >8 scoreable glomeruli were available from 27 subjects who constituted the Biopsy Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fostamatinib 150 mg | Fostamatinib 100 mg | Placebo | Total
Number analyzed (Participants) | 25 | 26 | 25 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 25 | 25 | 72
  >=65 years | 3 | 1 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (14.8) | 42.3 (14.1) | 40.6 (11.6) | 42.0 (40.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 13 | 40
  Male | 12 | 12 | 12 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | NA — Not collected | NA — Not collected | NA — Not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian | 11 | 6 | 6 | 23
  Native Hawaiian or Other Pacific Islander | NA — Not collected | NA — Not collected | NA — Not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American | 1 | 1 | 0 | 2
  White | 13 | 19 | 19 | 51
  More than one race | NA — Not collected | NA — Not collected | NA — Not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | NA — Not collected | NA — Not collected | NA — Not collected | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Mean Change of Proteinuria as Measured by Spot Urine Protein/Creatinine Ratio (sPCR) at Week 24
Description: Mean change from Baseline (Visit 2) of proteinuria as measured by the spot Protein-Creatinine Ratio (sPCR) at 24 weeks (Visit 9) for the ITT Population
Time Frame: Baseline to 24 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/g
Arm/Group | Fostamatinib 150 mg | Fostamatinib 100 mg | Placebo
Number analyzed (Participants) | 25 | 26 | 25
mg/g | -157.5 (345.6) | -577.2 (335.7) | -177.4 (342.4)
Statistical Analysis 1: Comparison: Fostamatinib 150 mg vs Placebo; Test type: Superiority; p = 0.97, ANCOVA; Mean Difference (Final Values) = 19.9, 95% CI 2-sided [-910.6 to 950.5]
Statistical Analysis 2: Comparison: Fostamatinib 100 mg vs Placebo; Test type: Superiority; p = 0.40, ANCOVA; Mean Difference (Final Values) = -399.7, 95% CI 2-sided [-1320.8 to 521.3]

2. Secondary Outcome: Mean Change From Pre-treatment to Post-treatment in Mesangial Hypercellularity (M) on Renal Biopsies.
Description: Mean change from pre-treatment to post-treatment in mesangial hypercellularity on renal biopsies. Using the Oxford Classification of IgA Nepthropathy (IgAN), biopsy specimens with a minimum of 8 glomeruli, mesangial hypercellularity (M), endocapillary hypercellularity (E), segmental sclerosis (S), and interstitial fibrosis/tubular atrophy (T) lesions are scored for assessing histologic findings in IgAN.
  M = the mean score based on Oxford Classification system score is based on total count of mesangial cells for all glomeruli (count of <4=0 score, 4 to 5=1, 6 to 7=2, ≥8=3). A decrease in score equates to improvement from IgAN disease.
Time Frame: Baseline to Week 24
Population: Analysis population includes only subjects with both pre-treatment and post-treatment biopsies collected.
Measure: Least Squares Mean (Standard Error); unit: mesangial hypercellularity score
Units Other Than Participants: renal biopsy samples
Arm/Group | Fostamatinib 150 mg | Fostamatinib 100 mg | Placebo
Number analyzed (Participants) | 3 | 13 | 11
Number analyzed (renal biopsy samples) | 6 | 26 | 22
mesangial hypercellularity score | -0.3 (1.6) | -0.2 (0.1) | -0.1 (0.1)

3. Secondary Outcome: Percentage of Subjects With ≥50% Reduction in sPCR From Baseline (Visit 2) at Week 24 (Visit 9).
Description: Percentage of subjects with ≥50% reduction in sPCR from Baseline (Visit 2) at Week 24 (Visit 9)
Time Frame: Baseline to Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib 150 mg | Fostamatinib 100 mg | Placebo
Number analyzed (Participants) | 25 | 26 | 25
Participants | 5 | 8 | 4

4. Secondary Outcome: Percentage of Subjects With ≥ 30% Reduction in Proteinuria From Baseline (Visit 2) at 24 Weeks (Visit 9).
Description: Percentage of subjects with ≥ 30% reduction in proteinuria from Baseline (Visit 2) at 24 weeks (Visit 9).
Time Frame: Baseline to Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib 150 mg | Fostamatinib 100 mg | Placebo
Number analyzed (Participants) | 25 | 26 | 25
Participants | 8 | 12 | 8

5. Secondary Outcome: Mean Change From Pre-treatment to Post-treatment in Percentage of Glomeruli With Endocapillary Hypercellularity (E) on Renal Biopsies.
Description: Mean change from pre-treatment to post-treatment in mesangial hypercellularity on renal biopsies. Using the Oxford Classification of IgA Nepthropathy (IgAN), biopsy specimens with a minimum of 8 glomeruli, mesangial hypercellularity (M), endocapillary hypercellularity (E), segmental sclerosis (S), and interstitial fibrosis/tubular atrophy (T) lesions are scored for assessing histologic findings in IgAN.
  E = Percentage of glomeruli eypercellularity due to increased number of cells within glomerular capillary lumina causing narrowing of the lumina. A decrease in score equates to improvement from IgAN disease.
Time Frame: Baseline to Week 24
Population: Analysis population includes only subjects with both pre-treatment and post-treatment biopsies collected.
Measure: Least Squares Mean (Standard Error); unit: Percentage of glomeruli
Units Other Than Participants: renal biopsy samples
Arm/Group | Fostamatinib 150 mg | Fostamatinib 100 mg | Placebo
Number analyzed (Participants) | 3 | 13 | 11
Number analyzed (renal biopsy samples) | 6 | 26 | 22
Percentage of glomeruli | -3.1 (3.2) | -4.0 (1.5) | -5.4 (1.7)

6. Secondary Outcome: Mean Change From Pre-treatment to Post-treatment in Percentage of Glomeruli With Segmental Sclerosis/Adhesion (S) on Renal Biopsies.
Description: Mean change from pre-treatment to post-treatment in mesangial hypercellularity on renal biopsies. Using the Oxford Classification of IgA Nepthropathy (IgAN), biopsy specimens with a minimum of 8 glomeruli, mesangial hypercellularity (M), endocapillary hypercellularity (E), segmental sclerosis (S), and interstitial fibrosis/tubular atrophy (T) lesions are scored for assessing histologic findings in IgAN.
  S = Percentage of any amount of the tuft involved in sclerosis, but not involving the whole tuft or the presence of an adhesion in each glomeruli. A decrease in score equates to improvement from IgAN disease.
Time Frame: Baseline to Week 24
Population: Analysis population includes only subjects with both pre-treatment and post-treatment biopsies collected.
Measure: Least Squares Mean (Standard Error); unit: Percentage of glomeruli
Units Other Than Participants: renal biopsy samples
Arm/Group | Fostamatinib 150 mg | Fostamatinib 100 mg | Placebo
Number analyzed (Participants) | 3 | 13 | 11
Number analyzed (renal biopsy samples) | 6 | 26 | 22
Percentage of glomeruli | -4.4 (7.8) | -6.8 (3.6) | -0.8 (3.9)

7. Secondary Outcome: Mean Change From Pre-treatment to Post-treatment in Percentage of Glomeruli With Global Glomerulosclerosis Score on Renal Biopsies.
Description: Mean change from pre-treatment to post-treatment in mesangial hypercellularity on renal biopsies. Using the Oxford Classification of IgA Nepthropathy (IgAN), biopsy specimens with a minimum of 8 glomeruli, mesangial hypercellularity (M), endocapillary hypercellularity (E), segmental sclerosis (S), and interstitial fibrosis/tubular atrophy (T) lesions are scored for assessing histologic findings in IgAN.
  Percentage of any amount of the tuft involved in sclerosis, but not involving the whole tuft or the presence of an adhesion in each glomeruli. A decrease in score equates to improvement from IgAN disease.
Time Frame: Baseline to Week 24
Population: Analysis population includes only subjects with both pre-treatment and post-treatment biopsies collected.
Measure: Least Squares Mean (Standard Error); unit: Percentage of glomeruli
Units Other Than Participants: renal biopsy samples
Arm/Group | Fostamatinib 150 mg | Fostamatinib 100 mg | Placebo
Number analyzed (Participants) | 3 | 13 | 11
Number analyzed (renal biopsy samples) | 6 | 26 | 22
Percentage of glomeruli | -11.9 (10.1) | 8.34 (4.8) | 0.5 (5.2)

8. Secondary Outcome: Mean Change From Pre-treatment to Post-treatment in Percentage of Glomeruli With Tubulointerstitial Scarring (T) on Renal Biopsies.
Description: Mean change from pre-treatment to post-treatment in mesangial hypercellularity on renal biopsies. Using the Oxford Classification of IgA Nepthropathy (IgAN), biopsy specimens with a minimum of 8 glomeruli, mesangial hypercellularity (M), endocapillary hypercellularity (E), segmental sclerosis (S), and interstitial fibrosis/tubular atrophy (T) lesions are scored for assessing histologic findings in IgAN.
  T= Percentage of cortical area involved by the tubular atrophy or interstitial fibrosis, whichever is greater. A decrease in score equates to improvement from IgAN disease.
Time Frame: Baseline to Week 24
Population: Analysis population includes only subjects with both pre-treatment and post-treatment biopsies collected.
Measure: Least Squares Mean (Standard Error); unit: Percentage of glomeruli
Units Other Than Participants: renal biopsy samples
Arm/Group | Fostamatinib 150 mg | Fostamatinib 100 mg | Placebo
Number analyzed (Participants) | 3 | 13 | 11
Number analyzed (renal biopsy samples) | 6 | 26 | 22
Percentage of glomeruli | -7.4 (9.7) | 4.4 (4.6) | -1.7 (5.0)

9. Secondary Outcome: Mean Change From Pre-treatment to Post-treatment in Percentage of Glomeruli With Cellular/Fibrocellular Crescent Score on Renal Biopsies.
Description: Mean change from pre-treatment to post-treatment in cellular/fibrocellular crescent score on renal biopsies. Biopsy specimens with a minimum of 8 glomeruli, mesangial hypercellularity (M), segmental sclerosis (S), and interstitial fibrosis/tubular atrophy (T) lesions are scored using the Oxford Classification of IgA nepthropathy (IgAN) system for assessing histologic findings in IgAN.
Time Frame: Baseline to Week 24
Population: Analysis population includes only subjects with both pre-treatment and post-treatment biopsies collected.
Measure: Least Squares Mean (Standard Error); unit: Percentage of glomeruli
Units Other Than Participants: renal biopsy samples
Arm/Group | Fostamatinib 150 mg | Fostamatinib 100 mg | Placebo
Number analyzed (Participants) | 3 | 13 | 11
Number analyzed (renal biopsy samples) | 6 | 26 | 22
Percentage of glomeruli | 2.3 (1.6) | -1.5 (0.8) | -0.4 (0.8)

10. Secondary Outcome: Mean Change From Baseline (Visit 2) of eGFR at 12 Weeks (Visit 7).
Description: Mean change from Baseline (Visit 2) of eGFR at 12 weeks (Visit 7).
Time Frame: Baseline to Week 12
Population: Analysis population includes only subjects who completed visits through Week 12.
Measure: Least Squares Mean (Standard Error); unit: eGFR (mL/min/1.73 m2)
Arm/Group | Fostamatinib 150 mg | Fostamatinib 100 mg | Placebo
Number analyzed (Participants) | 22 | 25 | 25
eGFR (mL/min/1.73 m2) | -2.0 (2.1) | 2.1 (1.9) | 1.4 (2.0)

11. Secondary Outcome: Mean Change From Baseline (Visit 2) of eGFR at 24 Weeks (Visit 9).
Description: Mean change from Baseline (Visit 2) of eGFR at 24 weeks (Visit 9).
Time Frame: Baseline to Week 24
Measure: Least Squares Mean (Standard Error); unit: eGFR (mL/min/1.73 m2)
Arm/Group | Fostamatinib 150 mg | Fostamatinib 100 mg | Placebo
Number analyzed (Participants) | 21 | 24 | 24
eGFR (mL/min/1.73 m2) | -0.9 (1.9) | 2.0 (1.8) | -0.2 (1.8)

12. Secondary Outcome: Mean Change From Baseline (Visit 2) of Proteinuria at 12 Weeks (Visit 7).
Description: Mean change from Baseline (Visit 2) of proteinuria at 12 weeks (Visit 7).
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: mg/g
Arm/Group | Fostamatinib 150 mg | Fostamatinib 100 mg | Placebo
Number analyzed (Participants) | 25 | 26 | 25
mg/g | -293.1 (202.0) | -529.2 (196.4) | -328.3 (199.9)

13. Secondary Outcome: Percentage of Subjects With sPCR <50 mg/mmol (500 mg/g) at 12 Weeks (Visit 7).
Description: Percentage of subjects with sPCR <50 mg/mmol (500 mg/g) at 12 weeks (Visit 7).
Time Frame: Baseline to Week 12
Measure: Number; unit: percentage of subjects
Arm/Group | Fostamatinib 150 mg | Fostamatinib 100 mg | Placebo
Number analyzed (Participants) | 25 | 26 | 25
percentage of subjects | 9 | 16 | 12

14. Secondary Outcome: Shift in Haematuria (Dipstick Test) From Baseline (Visit 2) at 12 Weeks (Visit 7).
Description: Shift in haematuria (dipstick test) from Baseline (Visit 2) at 12 weeks (Visit 7).
Time Frame: Baseline to Week 12
Measure: Number; unit: subjects
Arm/Group | Fostamatinib 150 mg | Fostamatinib 100 mg | Placebo
Number analyzed (Participants) | 25 | 26 | 25
subjects
  Increased | 1 | 0 | 0
  Same/Unchanged | 13 | 21 | 21
  Decreased | 8 | 4 | 4

15. Secondary Outcome: Shift in Haematuria (Dipstick Test) From Baseline (Visit 2) at 24 Weeks (Visit 9).
Description: Shift in haematuria (dipstick test) from Baseline (Visit 2) at 24 weeks (Visit 9).
Time Frame: Baseline to Week 24
Measure: Number; unit: subjects
Arm/Group | Fostamatinib 150 mg | Fostamatinib 100 mg | Placebo
Number analyzed (Participants) | 25 | 26 | 25
subjects
  Increased | 1 | 1 | 0
  Same/Unchanged | 14 | 15 | 19
  Decreased | 6 | 8 | 5

ADVERSE EVENTS:
Time Frame: The AE reporting period begins with the first dose of study drug and ends with the final study (follow-up) visit. AEs that occur between the time of consent and first dose of study drug will be reported as Medical History. If an SAE is present at the follow-up visit (Week 26, Visit 10) or final visit for subjects receiving extended treatment it was followed to resolution or stabilization unless the subject is lost to follow-up.
Arm/Group | Fostamatinib 150 mg | Fostamatinib 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/25 | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/25 | 2/26 | 2/25
Other Adverse Events (participants affected / at risk) | 24/25 | 22/26 | 21/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fostamatinib 150 mg (N=25) | Fostamatinib 100 mg (N=26) | Placebo (N=25)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post Procedural Haematuria (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Peptic Ulcer Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatic Enzyme Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fostamatinib 150 mg (N=25) | Fostamatinib 100 mg (N=26) | Placebo (N=25)
Diarrhoea (Gastrointestinal disorders) | 7 | 9 | 7
Nausea (Gastrointestinal disorders) | 5 | 6 | 3
Vomiting (Gastrointestinal disorders) | 4 | 3 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 3 | 1
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 4 | 1 | 7
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 1 | 5
Urinary Tract Infection (Infections and infestations) | 3 | 1 | 1
Alanine Aminotransferase Increased (Investigations) | 2 | 3 | 1
Aspartate Aminotransferase Increased (Investigations) | 1 | 2 | 1
Headache (Nervous system disorders) | 5 | 3 | 1
Dizziness (Nervous system disorders) | 1 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Hypertension (Vascular disorders) | 3 | 4 | 1
Gout (Metabolism and nutrition disorders) | 2 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/38/NCT02112838/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT02112838/SAP_001.pdf